CLINICAL TRIAL: NCT02513277
Title: Screening for Glucose Intolerance and Development of a Lifestyle Education Programme for Prevention of Type 2 Diabetes in a Population With Learning Disabilities
Brief Title: Diabetes Screening & Prevention for People With Learning (Intellectual) Disabilities:STOP Diabetes Study
Status: Completed | Type: Observational
Sponsor: University of Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: 0341; RP-PG-1209-10057 (Other Grant/Funding Number: NIHR Programme Grant for Applied Research)
Record Dates: First submitted 2015-07-29; First posted 2015-07-31 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2015-07

CONDITIONS: Diabetes Mellitus, Type 2; Prediabetic State; Intellectual Disability
Keywords: type 2 diabetes; impaired glucose regulation; intellectual disability; learning disability; screening; prevention; lifestyle education
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Prediabetic State; Intellectual Disability; Learning Disabilities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No

SUMMARY:
People with learning (intellectual) disabilities have more health problems than the rest of the population; they are less likely to access help and have lifestyles that may increase their risk of getting diabetes (for example, poor diet and lack of physical activity). People with learning disabilities may also be prescribed drugs or have certain medical conditions (such as Down's syndrome) which can make their chances of getting diabetes greater.

Diabetes is a long-term condition, which can cause damage to the eyes, heart, kidneys, nerves and feet. Impaired glucose regulation happens when sugar levels in the blood are higher than normal but are not high enough to be diagnosed with diabetes. People with impaired glucose regulation are more likely to develop diabetes, heart disease and stroke in the future. If people with impaired glucose regulation make changes to their lifestyle (diet and exercise) they can prevent or delay getting diabetes.

The aim of this study is to screen people with learning disabilities for diabetes and impaired glucose regulation. The investigators also want to find out the best way to give people with learning disabilities some education around healthy lifestyles (for example, eating and exercise) to help with prevention of diabetes and cardiovascular disease. Therefore, the investigators also aim to develop a lifestyle education programme that is suitable for use in this population and test whether it is feasible and acceptable.

DETAILED DESCRIPTION:
Background -Adults with learning (intellectual) disabilities tend to have more health problems than the general population and are less likely to access help. Additionally, evidence suggests that due to a combination of lifestyle factors (e.g. poor diet, lack of physical activity), associated medical problems, and certain types of prescribed medication, people with learning disabilities may be at increased risk of developing type 2 diabetes and cardiovascular disease. Our overall aim is to undertake a programme of research that improves our knowledge and understanding of screening for impaired glucose regulation and type 2 diabetes in a population with learning disabilities, and to develop a lifestyle education programme for prevention of type 2 diabetes that is suitable for use in this population.

SCREENING PROGRAMME

Aim - The main programme of work consists of a large diabetes screening programme. The primary aim of the screening study is to evaluate the feasibility and clinical and cost effectiveness of a screening programme for identifying undiagnosed type 2 diabetes and impaired glucose regulation that is suitable for use in a population with learning disabilities.

Methods - A variety of approaches will be used to recruit people to the screening study: General practices will be approached first for participation in this study. If the practice does not agree, then the investigators will seek to approach eligible people on the Leicestershire Learning Disabilities Register. Learning disabilities consultants will also approach people face to face when attending for outpatient clinic appointments. Additionally, if individuals with learning disabilities (and/or their carer) contact the STOP Diabetes team to express an interest in the study, they will be given an invitation.

* Volunteers will be asked to attend an appointment(s) where consent will be obtained and biomedical and demographic data collected. The consent process and data collection will be staged and people may need to attend between one to three appointments to complete.
* People who are found to have type 2 diabetes or impaired glucose regulation will be asked to see their GP for care.
* At every stage, reasonable adjustments will be made to take into account people's communication needs and decision making capacity. This may include involving a carer or a

DEVELOPMENT AND TESTING OF A STRUCTURED EDUCATION PROGRAMME

The aims of additional work being carried out alongside the screening study are to: (1) develop a lifestyle education programme to meet the needs of a population with learning disabilities and impaired glucose regulation or high risk of diabetes; (2) assess the feasibility of collecting outcome measures for participants with learning disabilities before and 3-months after they attend the education programme.

Methods - People approached to take part will be people who took part in the screening study and (1) gave their consent to be approached to take part in further phases of the research programme, and (2) were found to be at increased risk of developing diabetes according to their screening results.

Qualitative Interviews to inform curriculum development:

* Interviews will be conducted with a sample of people with mild/moderate learning disabilities, their carers and healthcare professionals. Findings from the interviews will help inform development of an initial curriculum and education program.

Delivery of initial curriculum and obtaining feedback:

* As part of the development work the education programme will be piloted with at least two groups of 6 - 8 people plus carers. Feedback will be collected from some of the people who attend the education sessions and any necessary changes made to the curriculum. These cycles of piloting, collecting feedback and modifying the programme will be repeated until the education programme developed is "fit for purpose".

Delivery of programme with collection of before and after measures:

* Following initial development, testing and refinement of the curriculum, the education programme will be delivered with another sample of participants and the feasibility of collecting pre and post intervention outcome measures will be tested. The investigators anticipate delivering the programme to up to two groups of 6 - 8 people plus carers. Data will be collected at baseline and 3-months (12 weeks) following delivery of the final education session. Data and may include: physical activity and sedentary behaviour (as measured by accelerometer); body weight, BMI, waist circumference, blood pressure and dietary intake (fruit and vegetables). Uptake of the education programme (attendance) and retention at 3-months follow-up will also be explored. This phase will be subject to modification depending on the findings from prior iterations and any problems encountered.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer has a confirmed learning disability (permanent intellectual impairment);
* Registered with a general practice in Leicester, Leicestershire or Rutland, UK;
* Participant and/or carer has sufficient English language skills to enable fully informed consent to be obtained.

Exclusion Criteria:

* Confirmed diagnosis of Type 2 diabetes or Type 1 Diabetes;
* Malignancy or terminal illness;
* Pregnancy or breast feeding;
* Severe systemic disease that may interfere with measurement and interpretation of HbA1c.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults with a learning (intellectual) disability who are live in Leicester, Leicestershire or Rutland, UK;
Sampling Method: Non-Probability Sample
Enrollment: 930 (Actual)
Dates: Start 2013-02; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Glycosylated haemoglobin (HbA1c) | Baseline screening appointment
  Identification of type 2 diabetes, impaired glucose regulation, or normal glucose regulation
Plasma glucose | Baseline screening appointment
  Identification of type 2 diabetes, impaired glucose regulation, or normal glucose regulation

SECONDARY OUTCOMES:
Physical activity levels (including sedentary behaviour) | Baseline screening appointment
  measured by accelerometer - only for a small sub-group
Obesity levels | Baseline screening appointment
  body mass index and waist size
Blood pressure | Baseline screening appointment
  systolic and diastolic
Lipids levels | Baseline screening appointment
  total cholesterol, LDL, HDL, triglycerides
Dietary/nutritional intake | Baseline screening appointment
  food groups and fruit and vegetable intake
Cardiovascular risk | Baseline screening appointment
  Framingham risk score
Health related quality of life | Baseline screening appointment
  EQ-5D
Behavioural disorders | Baseline screening appointment
  Aberrant Behaviour Checklist
Psychiatric disorders | Baseline screening appointment
  PAS-ADD checklist
Depression | Baseline screening appointment
  Glasgow Depression Scale and Carer Supplement

CONTACTS AND LOCATIONS:
Overall Officials: Prof Kamlesh Khunti, PhD, FRCGP, Principal Investigator — Diabetes Research Centre, University of Leicester; Prof Sabyasachi Bhaumik, FRCPsych, Principal Investigator — Learning Disability Service, Leicester Partnership NHS Trust
Locations (1):
- Diabetes Research Centre, University of Leicester, Leicester, United Kingdom